CLINICAL TRIAL: NCT04231370
Title: Combination of Lenalidomide and Sintilimab for Patients With Relapsed/Refractory NK/T-cell Lymphoma Who Failed Pegaspargase-based Regimens: a Single Arm, Open, Phase II Study
Brief Title: Lenalidomide and Sintilimab for Relapsed/Refractory NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, JING-WEN WANG, Professor of Department of Hematology, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRhos-ENKTCL-1
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: NK/T Cell Lymphoma Nos
Keywords: pegaspargase; sintilimab; PD-1; lenalidomide; relapsed/refractory
MeSH Terms: conditions — Recurrence | interventions — sintilimab; spartalizumab; Lenalidomide; Immunomodulating Agents

STUDY DESIGN:
Intervention Model Description: treatment with lenalidomide in combination with sintilimab for relapsed/refractory ENKTCL patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Sintilimab, 200mg, iv day1 Lenalidomide, 25mg/d, oral, day 1-14 repeated every 3 weeks
  Interventions: Drug: Sintilimab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Sintilimab — Sintilimab, 200mg, iv day1
  Other Names: anti-PD-1-antibody
Drug: Lenalidomide — 25mg/d oral d1-14
  Other Names: IMids

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Sintilimab in combination with lenalidomide in the treatment of Relapsed/Refractory NK/T-cell lymphoma patients who failed pegaspargase-based regimens.

DETAILED DESCRIPTION:
Pegaspargase is the backbone of treatment for NK/T-cell lymphoma (ENKTCL), and patients with ENKTCL who failed pegaspargase-based regimens have extremely poor survival outcomes. Previous study has confirmed the efficacy of anti-PD-1 antibodies (including pembrolizumab or sintilimab). Constitutive activation of NF-kB pathway has been demonstrated to be involved in the development of ENKTCL and plays critical role in therapy resistance. Lenalidomide, an immuno-modulatory drug, has been found to inhibit NF-kB pathway, and synergize with anti-PD-1 antibody in the treatment of multiple myeloma. Thus, we hypothesize that the combination of lenalidomide and sintilimab will further deepen the remission status and benefit patients who failed pegaspargase-based regimens.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology and immunohistochemistry confirmed diagnosis of NK/T-cell lymphoma according to WHO 2016 criteria.
* Previously treated with pegaspargase-based regimens (refractory or relapsed after initial remission).
* PET/CT or CT/MRI with at least one objectively evaluable lesion.
* General status ECOG score 0-3 points.
* The laboratory test within 1 week before enrollment meets the following conditions:

Blood routine: Hb>80g/L, PLT>50×10（9）/L. Liver function: ALT, AST, TBIL ≤ 2 times the upper limit of normal. Renal function: Cr is normal. Coagulation : plasma fibrinogen ≥ 1.0g / L. Cardiac function: LVEF≥50%, ECG does not suggest any acute myocardial infarction, arrhythmia or atrioventricular conduction above I Blocking.

* Sign the informed consent form.
* Voluntary compliance with research protocols, follow-up plans, laboratory and auxiliary examinations.

Exclusion Criteria:

* Patients with a history of pancreatitis.
* Active infection requires ICU treatment.
* Concomitant HIV infection or active infection with HBV, HCV. Patients who are infected with HBV but not active hepatitis at the same time are not excluded.
* Serious complications such as fulminant DIC.
* Significant organ dysfunction: such as respiratory failure, NYHA classification ≥ 2 chronic congestive heart failure, decompensation Hepatic or renal insufficiency, high blood pressure and diabetes that cannot be controlled despite active treatment, and cerebral vascular thrombosis or hemorrhagic time within the past 6 months.
* Pregnant and lactating women.
* Had a history of autoimmune diseases, and disease was active in the last 6 months, and was still taking oral immunosuppression in the past three months.
* Those who were known to be allergic to drugs in the study regimen.
* Patients with other tumors who require surgery or chemotherapy within 6 months.
* Other experimental drugs are being used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of complete response | 24 weeks ±7 days
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria

SECONDARY OUTCOMES:
Rate of overall response | 24 weeks ±7 days
  evaluated by PET-CT and MRI, according to Lugano 2014 criteria
1-year progression free survival rate | up to 1year after enrollment
  time from date of enrollment to date of disease progression, death of any reason, whichever comes first
1-year overall survival rate | up to 1year after enrollment
  time from date of enrollment to date of death of any reason
safety profiles | up to 1year after enrollment
  according to CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jing-wen Wang, M.D., Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
All the data in the trial can be shared upon request to the PI.